CLINICAL TRIAL: NCT03048617
Title: A Prospective Observational Study of Patients With Primary Mitochondrial Disease (SPIMM-300)
Brief Title: An Observational Study of Patients With Primary Mitochondrial Disease (SPIMM-300)
Acronym: RePOWER
Status: Completed | Type: Observational
Sponsor: Stealth BioTherapeutics Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SPIMM-300
Record Dates: First submitted 2017-02-03; First posted 2017-02-09 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Primary Mitochondrial Disease
Keywords: Primary Mitochondrial Disease; Stealth; Myopathy; exercise intolerance; muscle pain; Mitochondrial Myopathy; Primary Mitochondrial Myopathy
MeSH Terms: conditions — Muscular Diseases; Myalgia; Mitochondrial Myopathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is an observational study of patients with Primary Mitochondrial Disease with either signs or symptoms suggestive of myopathy. The Investigator will identify potential patients through existing medical records and one on-site visit.

DETAILED DESCRIPTION:
An observational study of patients with presumed Primary Mitochondrial Disease designed to better characterize and correlate symptoms and signs of myopathy and genetic test results and the use of commonly prescribed treatments. The study will help define and identify a subject population for a future trial of an investigational product to treat primary mitochondrial disease associated with signs and symptoms of myopathy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide a signed informed consent form (ICF) prior to participation in any-trial related procedures
* Patient has clinical presentation of PMD with either signs or symptoms suggestive of myopathy
* Patient is ambulatory and able to attempt 6MWT

Exclusion Criteria:

* Patient has symptoms of PMD due to secondary mitochondrial dysfunction
* Patient has had prior exposure to elamipretide
* Patient does not have the cognitive capacity to understand and complete all study assessments
* Patient has a medical history of severe renal impairment
* History of active alcoholism or drug addiction during the year before enrollment

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with clinical presentation of PMD with either signs or symptoms suggestive of myopathy
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2018-08-02 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Assess the relationship of genotype to phenotype in patients with Primary Mitochondrial Disease | 1 year
Compare local and regional differences in standard of care and management of patients with Primary Mitochondrial Disease | 1 year

SECONDARY OUTCOMES:
Compare local and regional differences in genetic testing methodologies for Primary Mitochondrial Disease | 1 year

CONTACTS AND LOCATIONS:
Locations (33):
- United States (13):
  - University of California San Diego, La Jolla, California
  - Stanford Universtity, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center, Houston, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
- Australia (2):
  - Calvary Health Care Bethlehem, Caulfield South, Victoria
  - Royal North Shore Hospital, St Leonards
- Canada (3):
  - University of Calgary Metabolic Disease Clinica, Calgary, Alberta
  - McMaster University Medical Center, Hamilton, Ontario
  - Adult Metabolic Diseases Clinic, Vancouver
- University of Copenhagen, Copenhagen, Denmark
- Germany (2):
  - Klinikim der Universitat Muchen, Friedrich-Baur Institute, Munich, Bavaria
  - University Hospital of Bonn, Bonn
- Institute of Genomic Medicine and Rare Disorders, Budapest, Hungary
- Italy (7):
  - IRCCS Institute of Neurological Sciences of Bolgna, Bellaria Hospital, Bologna
  - ASST Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero Universitaria Policlinico G. Martino, Messina
  - Istituto Nazionale Neurologico Carlo Besta, Milan
  - Istituto di Neurologia, Fondazione Policlinico Universitario A. Gemelli, Roma
  - Dipartimento Ambientale di Neuroscienze, Roma
  - Ospedale Pediatrico Bambin Gesu, Roma
- Spain (2):
  - Hospital Universitario 12 de Octubre, Madrid
  - Neurology Department Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (2):
  - MRC Centre for Neuromuscular Diseases, London
  - Royal Victoria Infirmary, Newcastle upon Tyne